CLINICAL TRIAL: NCT02802436
Title: The Impact of a Known Bioactive Agent on the Resolution of Alveolar Socket Preservation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Administrative changes precluded enrollment.
Sponsor: Boston University (Other)
Collaborators: OsteoHealth (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H34663
Record Dates: First submitted 2016-06-07; First posted 2016-06-16 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Healing of Extraction Socket
MeSH Terms: interventions — socket graft

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Extraction with socket graft and GEM21 (Experimental): Intervention - Extraction will be done as usual standard of care to preserve socket walls. Graft material (mineralized cortical/cancellous Bone Powder 250-1000µ) will be used, site will be filled slightly below marginal bone level (1mm). Test site (active arm) will be injected with Bioactive Agent (PDGF - Platelet derived growth factor). At 3 levels apical 1/3rd, middle 1/3rd and coronal 1/3rd.
  Bioactive agent - GEM21S (Growth factor enhanced matrix) Dosage - one cup containing 0.5 cc of ß-TCP particles (0.25 to 1.0 mm); and one syringe containing a solution of 0.5 mL rhPDGF-BB (0.3 mg/mL)
  Interventions: Procedure: Extraction with socket graft
- Extraction with socket graft (Other): Extraction will be done as usual standard of care to preserve socket walls. Graft material (mineralized cortical/cancellous Bone Powder 250-1000µ) will be used, site will be filled slightly below marginal bone level (1mm). Normal saline will be used and no growth factor to maintain the volume in control sites
  Interventions: Procedure: Extraction with socket graft

INTERVENTIONS:
Procedure: Extraction with socket graft — Extraction will be done as usual standard of care to preserve socket walls. Sockets will be measured at all 4 line angles for depth with the same periodontal probe, Buccal-Lingual dimension will be measured prior to graft placement. Graft material (mineralized cortical/cancellous Bone Powder 250-1000µ) will be used for both sites. Volume of graft used will be recorded. Both sites will be filled slightly below marginal bone level (1mm). Test site will be injected with Bioactive Agent. At 3 levels apical 1/3rd, middle 1/3rd and coronal 1/3rd. Control site will be injected with saline (or vehicle) at same levels. Occlusal orifice will be closed with Collagen plug adjusted for depth to meet free gingival margins and then sutured with 4-0 PGA (Vicryl)

SUMMARY:
The advent of endosseous implant restoration has driven an increasing need for alveolar bone preservation and/or augmentation strategies. Investigations have explored the physical scaffold effects of a wide variety of bone graft materials with each graft material offering a more or less attractive surface for bone deposition. The seeding of these scaffolds with biologically active material seeks to enhance the "osteoconductive" effect by influencing the temporal or sequential steps which result in the desired end product-new bone.

Alveolar socket grafts are a common example of these preservation techniques. They are an accepted procedure to maximize the retention of alveolar bone post extraction. They appear to act as a passive scaffold for clot retention and subsequent bone regeneration.

The current pilot research project explores addition of a known Bioactive Agent: Platelet Derived Growth Factor (PDGF) to test its impact on healing responses. Histomorphometric assessments will be utilized on microscopic slide material derived from cores trephined as the initial step in the preparation for placement of endosseous dental implants. Outcomes measured will include:

Clinical observation of healing response

Microscopic measures will be

* Measures of residual graft material
* New bone formation and new bone contact area with graft
* Measures of vascular content
* Osteoclast count
* Qualitative measures of other marrow components (Cells and relative fiber/ fat content, liner cell characteristics.)

DETAILED DESCRIPTION:
The current pilot research project explores the addition of a known Bioactive Agent: Platelet Derived Growth Factor (PDGF) into the completed "socket graft" to test its impact on healing responses. Histomorphometric and qualitative assessments will be utilized on microscopic slide material derived from cores trephined as the initial step in the osteotomy preparation for placement of endosseous dental implants.

Design: Split mouth RCT (Randomized controlled trial) Graft Procedure: At time of extraction the site will be asked to rinse with 0.12% Chlorhexidine, and anesthetized with 2% lidocaine and 1/100,000 epinephrine. Extraction will be done as usual standard of care to preserve socket walls. Sites requiring socket wall repair at time of extraction will be excluded from study. Sockets will be measured at all 4 line angles for depth with the same periodontal probe, Buccal-Lingual dimension will be measured prior to graft placement. Graft material (mineralized cortical/cancellous Bone Powder 250-1000µ) will be used for both sites. Volume of graft used will be recorded. Both sites will be filled slightly below marginal bone level (1mm). Test site will be injected with Bioactive Agent. At 3 levels apical 1/3rd, middle 1/3rd and coronal 1/3rd. Control site will be injected with saline (or vehicle) at same levels. Occlusal orifice will be closed with Collagen plug adjusted for depth to meet free gingival margins and then sutured with 4-0 Polyglactin (Vicryl)

Post op care: Sites will be checked and photographed at 1 week, 2 weeks (sutures removed) and clinical photos taken to monitor clinical signs of inflammation and healing. A 3-month post op radiograph appointment will be made at the 2-week visit. Ct scan may be taken if prescribed by treatment plan/ prior to implant placement.

Implant/core acquisition at time of Implant placement: Clinical photographs will be taken. (Post graft radiograph already done at 3 months) Site will be opened with standard full thickness flap entry. After soft tissue reflection photo will be taken and implant site marked with a standardized round bur to ½ depth of bur (~ 0.5-1.0 mm). Sites requiring a 4, 5, or 6mm implant will have trephined core as first step in osteotomy (3.3mm OD-2-8mmID) Trephine will be centered over site mark and osteotomy and prepared to prescribed depth. The trephine core will be photographed with periodontal probe included for reference of length, apical end marked with India ink and then placed in 10% neutral buffered formalin (NBF) and labeled with patient name, date, record # and length of core. Details of implant placement will be recorded with size of implant and insertion torque in record.

Post-implant care: Standard of care post op sequence will be followed, once adequate healing period has elapsed healing cap that was screwed onto the implant is removed and replaced with appropriately shaped abutment. The entire procedure will be photographed and the usual post abutment radiograph will be taken at that time.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be selected from the pool of periodontal patients at BUSDM (Boston University School of Dental Medicine) who have been treatment planned for at least two extractions which will be atleast one tooth apart in either arch (maxilla or mandible) followed by delayed 3-4 months dental implant placement.
* Subjects will be in age group 20-80 years of age.

Exclusion Criteria:

* Patients with known systemic disorders affecting bone Example - Osteoporosis, Diabetes Mellitus, Hyperthyroidism, Arthritis, smokers and pregnant women will be excluded.
* Untreated acute infections at the surgical site
* Untreated malignant neoplasm(s) at the surgical site
* Patients with a known hypersensitivity to any product component (ß-TCP = Tri calcium phosphate or rhPDGF-BB = Platelet derived growth factor)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10-03 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Implant/core acquisition at time of Implant placement | 3 months
  Site will be opened with standard full thickness flap entry. After soft tissue reflection photograph will be taken and implant site marked with a standardized round bur to ½ depth of bur (~ 0.5-1.0 mm). Sites requiring a 4, 5, or 6mm implant will have trephined core as first step in osteotomy (3.3mm OD-2-8mmID) Trephine will be centered over site mark and osteotomy and prepared to prescribed depth. The trephine core will be photographed with periodontal probe included for reference of length, apical end marked with India ink and then placed in 10% neutral buffered formalin (NBF) and labeled with patient name, date, record # and length of core. Details of implant placement will be recorded with size of implant and insertion torque in record.

CONTACTS AND LOCATIONS:
Overall Officials: Sunny K Tilwani, BDS, Principal Investigator — Boston University Dental School; Albert Price, DMD, Study Chair — Boston University Dental School
Locations (1):
- Henry M. Goldman School of Dental Medicine, Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Albrektsson T, Johansson C. Osteoinduction, osteoconduction and osseointegration. Eur Spine J. 2001 Oct;10 Suppl 2(Suppl 2):S96-101. doi: 10.1007/s005860100282. PMID 11716023
- [Result] Nevins M, Giannobile WV, McGuire MK, Kao RT, Mellonig JT, Hinrichs JE, McAllister BS, Murphy KS, McClain PK, Nevins ML, Paquette DW, Han TJ, Reddy MS, Lavin PT, Genco RJ, Lynch SE. Platelet-derived growth factor stimulates bone fill and rate of attachment level gain: results of a large multicenter randomized controlled trial. J Periodontol. 2005 Dec;76(12):2205-15. doi: 10.1902/jop.2005.76.12.2205. PMID 16332231
- [Result] Jayakumar A, Rajababu P, Rohini S, Butchibabu K, Naveen A, Reddy PK, Vidyasagar S, Satyanarayana D, Pavan Kumar S. Multi-centre, randomized clinical trial on the efficacy and safety of recombinant human platelet-derived growth factor with beta-tricalcium phosphate in human intra-osseous periodontal defects. J Clin Periodontol. 2011 Feb;38(2):163-72. doi: 10.1111/j.1600-051X.2010.01639.x. Epub 2010 Dec 6. PMID 21133980